CLINICAL TRIAL: NCT06883071
Title: Clinical Study on the Selection of Endoscopic Varicose Disconnection Strategy Based on Natural Portal Shunt with Portal Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaolong Zheng, Experimental researcher, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YAN2024-0545
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental)
  Interventions: Procedure: Endoscopic ultrasound (EUS)-guided spring plug combined with ECI
- Group B (Active Comparator)
  Interventions: Procedure: Titanium clip plus EUS-guided spring plug placement for flow limiting combined with ECI

INTERVENTIONS:
Procedure: Endoscopic ultrasound (EUS)-guided spring plug combined with ECI — Group A: Spring plug combined with ECI under the guidance of endoscopic ultrasound (EUS): Spring plug was placed to limit the flow of varicose veins by EUS, and then tissue glue was injected under EUS to block the varicose veins. Group B: Titanium clip plus EUS-guided spring plug placement to limit the flow combined with ECI: After partial titanium clip flow limitation under endoscopy, spring coil combined with tissue glue injection was placed in the varicose veins by judging the inflow and outflow tracts under the guidance of ultrasound (EUS).
  Arms: Group A
Procedure: Titanium clip plus EUS-guided spring plug placement for flow limiting combined with ECI — Group A: Spring plug combined with ECI under the guidance of endoscopic ultrasound (EUS): Spring plug was placed to limit the flow of varicose veins by EUS, and then tissue glue was injected under EUS to block the varicose veins. Group B: Titanium clip plus EUS-guided spring plug placement to limit the flow combined with ECI: After partial titanium clip flow limitation under endoscopy, spring coil combined with tissue glue injection was placed in the varicose veins by judging the inflow and outflow tracts under the guidance of ultrasound (EUS).
  Arms: Group B

SUMMARY:
Research content: This trial follows the randomized controlled study protocol to study the varicose vein elimination rate, amount of tissue glue used, rebleeding rate, complications, mortality, length of hospital stay, treatment costs, etc. of different endoscopic treatment methods for GV patients, and combines the correlation of factors such as etiology, liver function grade, and gender. So as to formulate the best treatment strategy for endoscopic treatment of GV patients.

Research objectives: By collecting case data, blood tests, gastroscopy reports, and CTP examination results of GV patients, endoscopic secondary prevention interruption surgery is performed on them. Compare the varicose vein elimination rate, amount of tissue glue used, rebleeding rate, complications, mortality, length of hospital stay, treatment costs, etc. of GV patients after endoscopic treatment, and evaluate the efficacy of different endoscopic treatment methods. At the same time, combined with factors such as etiology, liver function grade, and gender, formulate the best strategy for endoscopic interruption treatment of GV patients.

Key scientific issues to be addressed: a. Compare the efficacy of different endoscopic treatments for gastric varices with natural portosystemic shunts b. Provide a basis for strategic selection for endoscopic devascularization of gastric varices 5. Research methods, technical routes and schedule Research methods

1. Clinical trial registration All patients complied with the Declaration of Helsinki, and the study was reviewed and approved by the Ethics Committee of the Second Affiliated Hospital of Zhejiang University School of Medicine.
2. Patient inclusion and related examinations 32 patients with GV were included, with the following inclusion criteria: 1. Age ≥ 18 years; 2. History of liver cirrhosis and previous portal hypertension bleeding; 3. Endoscopic and abdominal CT assessment of IGV1 varicose veins and presence of SPSS; 4. Patients agreed to EUS treatment Exclusion criteria: 1. Previous treatment for portal hypertension bleeding (including endoscopy, intervention, and surgery); 2. Patients with critical illness, pregnant patients, immunodeficiency diseases (such as systemic lupus erythematosus), and mental illness; 3. Patients who refused endoscopic treatment
3. Implementation of the plan:

   All patients with complete hemodynamic characteristics of gastric varicose veins and stable vital signs were treated with endoscopic interruption of flow and signed a consent form for treatment; all patients were randomly divided into 2 groups (random table established), with 16 patients in each group. Group A: endoscopic ultrasound (EUS)-guided spring plug combined with ECI: Spring plug was placed to limit flow in varicose veins determined by EUS, and then tissue glue was injected under EUS to block varicose veins. Group B: Titanium clip plus EUS-guided spring plug flow limiting combined with ECI: After partial endoscopic titanium clip flow limiting, spring coils were placed in the varicose veins under ultrasound (EUS) guidance to determine the inflow and outflow tracts and to inject woven glue. Patients in both groups underwent CTP and gastroscopy follow-up at 1 month, 3 months, and 6 months after the initial treatment, and additional endoscopic treatment was performed if necessary; if bleeding occurred again during the period, timely treatment was given according to the condition (drugs, endoscopy, intervention or surgery); if other complications occurred, if they did not affect the study, the planned plan was continued.
4. Comparative analysis of results:

The postoperative bleeding rate of patients in the two groups after gastroscopy diagnosis and treatment was observed and compared (including a. short-term bleeding rate within 72 hours: hematemesis or black stool; systolic blood pressure decreased by >20 mmHg or heart rate increased by >20 times/min; in the absence of blood transfusion: hemoglobin decreased by >30 g/L; b. rebleeding: active bleeding occurred within 6 months; differences in hospitalization time and cost, as well as gender, age, etiology, basic liver function, etc. were further compared.)

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old; 2. History of liver cirrhosis and previous portal hypertension bleeding; 3. Endoscopic and abdominal CT evaluation of IGV1 varicose veins and the presence of SPSS; 4. The patient agrees to treatment under EUS

Exclusion Criteria:

* 1. Patients who have received treatment for portal hypertension bleeding (including endoscopy, intervention, and surgery) in the past; 2. Patients with critical illness, pregnant patients, immunodeficiency diseases (such as systemic lupus erythematosus), and mental illness; 3. Patients who refuse endoscopic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Observation and comparison of bleeding rates after gastroscopy in two groups | Gastroscopy follow-up was performed 1 month, 3 months, and 6 months after treatment.
  The bleeding rates after gastroscopy diagnosis and treatment were observed and compared between the two groups (including a. short-term bleeding rate within 72 hours: hematemesis or melena; systolic blood pressure decreased by >20 mmHg or heart rate increased by >20 times/min; in the absence of blood transfusion: hemoglobin decreased by >30 g/L; b. rebleeding: active bleeding within 6 months; differences in hospitalization time and cost, as well as gender, age, etiology, basic liver function, etc. were further compared).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol